CLINICAL TRIAL: NCT03871244
Title: Pilot Optimizing Transfusion Thresholds in Critically-ill Children With Anaemia (P-OpTTICCA): a Pilot Trial for a Large Pragmatic International Parallel Open-label Non-inferiority Randomised Controlled Trial.
Brief Title: Pilot Optimizing Transfusion Thresholds in Critically-ill Children With Anaemia
Acronym: P-OpTTICCA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); Hôpital Jeanne de Flandre (Unknown); NHS Blood and Transplant (Other Government)
Responsible Party: Principal Investigator, Jacques Lacroix, MD, FRCPC, Professor, Professor, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP-21-2019-2235
Record Dates: First submitted 2019-03-06; First posted 2019-03-12 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Anemia
Keywords: hemoglobin threshold; critically ill children; randomized controlled trial; red blood cell tranfusions
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: parallel open-label pragmatic non-inferiority randomised controlled trial (RCT)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restrictive arm (intervention) (Experimental): Less red blood cell transfusions. The protocol will require that no red blood cell transfusion be given unless the hemoglobin level is below or equal at 70 g per L.
  Interventions: Procedure: Less red blood cell transfusions
- Standard care arm (comparator) (Active Comparator): Clinical teams will follow their usual transfusion practices.
  Interventions: Procedure: More red blood cell transfusion (standard transfusion strategy in PICU)

INTERVENTIONS:
Procedure: Less red blood cell transfusions — The instructions given to caregivers will be to consider prescribing a red blood cell transfusion only if the hemoglobin level is ≤ 70 g per L.
  Other Names: Restrictive red blood cell transfusion strategy
  Arms: Restrictive arm (intervention)
Procedure: More red blood cell transfusion (standard transfusion strategy in PICU) — The instructions given to caregivers will be to prescribe a red blood cell transfusion according to their usual standard practice
  Arms: Standard care arm (comparator)

SUMMARY:
The Pilot Optimizing Transfusion Thresholds in Critically-ill Children with Anaemia (P-OpTTICCA) study is a pilot trial for a large pragmatic international parallel open-label non-inferiority randomised controlled trial. The primary outcome of the pilot study is feasibility.

DETAILED DESCRIPTION:
Patients in paediatric intensive care units (PICU) are among the main groups of transfusion recipients. Blood transfusions expose recipients to infectious and non-infectious serious hazards. Despite an increasing number of red blood cell (RBC) transfusion threshold randomised controlled trials (RCT) to date, only one large RCT, the Transfusion Requirement In PICU (TRIPICU) study (Lacroix. N Engl J Med 2007;356:1609-19) informs practice in PICU. This dearth of paediatric data was reiterated by a recent National Heart, Lung and Blood Institutes state of the art symposium. Despite being internally robust, the generalizability of TRIPICU has been questioned given that nearly 90% of critically ill children with haemoglobin (Hb) level ≤ 95 g/L were not enrolled for a range of pre-specified reasons including severity of illness, clinical instability and uncertain physician buy-in, thus threatening broader application of this critical knowledge into practice. Recent data and evidence summarised in systematic reviews support the need to explore the benefits and safety of Hb threshold ≤ 70 g/L for almost all critically ill children, not only those who would have been enrolled in TRIPICU.

We propose an international pilot study that will inform the design of a large pragmatic non-inferiority RCT (termed OpTTICCA) conceived to derive generalizable transfusion guidance for physicians.

Objectives of the pilot-RCT. Specific aims are to:

1. Establish the feasibility of enrolling ≥80% of eligible patients.
2. Document adherence to study intervention ≥80% (restrictive transfusion policy).
3. Assess the incidence rate of the primary outcome measure of the full RCT (new and progressive multiple organ dysfunction syndrome, which includes mortality).
4. Establish the feasibility of using routinely collected clinical information from electronic medical data monitoring system (eMDMS) to enhance cost-efficiency.

In the pilot-RCT, we will enrol 120 patients (20 to 40/site) in PICUs equipped with electronic medical data monitoring system (eMDMS). This trial builds on successful prior RCTs that involved international collaboration and funding (Canada, United Kingdom, France): TRIPICU, Age of Blood Evaluation (ABLE) (Lacroix. N Engl J Med 2015) and Age of Blood in Children in PICU (ABC-PICU study: Tucci et al. Trials 2018). The pilot-RCT will be considered as the vanguard phase of the full OpTTICCA RCT if no important design changes are required.

Expected results. This pilot-RCT will focus on feasibility parameters. It will explore whether we can 1) recruit a much broader eligible patient group, 2) assess protocol adherence, 3) assess the primary outcome measure, and 4) abstract most data electronically. A definitive trial will provide transfusion guidance for many important subgroups in whom evidence is presently lacking including children admitted with bone marrow failure, head injury, some cardiac disorders, and sepsis.

ELIGIBILITY:
Inclusion Criteria:

* 1. Hemoglobin concentration ≤ 95 g/L, while in PICU
* 2. Not already participating to a randomized controlled trial on hemoglobin threshold to guide red blood cell transfusion practice

Exclusion Criteria:

1. Post conception age ≤ 36 weeks or > 18 years at PICU entry
2. Refusal of consent by patient and/or parent
3. Uncorrected cyanotic cardiac disease, univentricular physiology
4. Sickle cell disease
5. Brain Death
6. Extracorporeal membrane oxygenation (ECMO)

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment: screening | One year
  Proportion of patients eligible for consent approached > 90%;
Recruitment: consent | One year
  Proportion of approached patients who decline consent < 20%,
Recruitment: enrolment | One year
  Recruitment: ≥ 2 patients randomized/site/week.

SECONDARY OUTCOMES:
Representativeness: exclusion | One year
  We recruit > 80% of patients who would have been excluded from TRIPICU (Lacroix et al. N Engl Med 2007).
Representativeness: opt-out | One year
  Proportion of dropout and lost to follow-up is expected to be < 2%.
Compliance | One year
  Proportion of RBC transfusions given with hemoglobin > 70 g/L in the restrictive arm (definition of non-compliance) is < 20%.
Separation | One year
  Post randomisation separation of hemoglobin concentration between both arms in the pilot-RCT is ≥ 10 g/L.
Suspension | One year
  Proportion of children wha are suspended is < 20%.
Data collection | One year
  Most data (> 80%) are abstracted directly from electronic medical data monitoring system.
Data entry | One year.
  Proportion of erroneous data entry is < 5%.
Outcomes | One year.
  Incidence rate of the primary outcome measure - new and progressive multiple organ dysfunction syndrome (NPMODS) - in the standard care arm of the pilot-trial is ≥ 20%.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Lacroix, Principal Investigator — St-Justine Hospital Center
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
The data of P-OpTTICCA will be integrated in the large trial if possible. This will not be possible if P-OpTTICCA shows that significant changes must be made to the research proposal of the full trial; then the data of participants of P-OpTTICCA will be merged to the data of the full trial using a meta-analysis strategy.

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Tucci M, Sarfatti A, Leteurtre S, Du Pont-Thibodeau G, Fontela P, Ray S, Stanworth SJ, Hebert PC, Roumeliotis N, Sauthier M, Spinella PC, Ducruet T, Jouvet P, Masse B, Robitaille N, Trottier H, Lacroix J; Canadian Critical Care Trials Group and the Groupe Francophone de Reanimation et d'Urgences Pediatriques. Pilot-Optimizing Transfusion Therapy in Critically Ill Children With Anemia: A Pilot Multicenter Electronic Health Record-Enabled Randomized Controlled Trial on Red Blood Cell Transfusion in Critically Ill Children. Pediatr Crit Care Med. 2025 Oct 1;26(10):e1218-e1230. doi: 10.1097/PCC.0000000000003822. Epub 2025 Sep 12. PMID 40938139
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836